CLINICAL TRIAL: NCT01681550
Title: Effect of Incretin-based Therapy Combined With Insulin on HbA1c, Hypoglycemia and Chronic Diabetic Complications in Type 2 Diabetic Patients
Brief Title: A Cohort Study of Incretin-based Therapy Combined With Insulin in Type 2 Diabetic Patients for 5 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, MD, Nagaoka Red Cross Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-Kamoi
Record Dates: First submitted 2012-09-02; First posted 2012-09-10 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Incretin theapy combined with insulin (Other)
  Interventions: Drug: Incretin-based therapy

INTERVENTIONS:
Drug: Incretin-based therapy

SUMMARY:
The use of dipeptidyl-peptidase 4 (DPP-4) inhibitors and glucagon like peptide 1 (GLP1) analogues for the treatment of diabetic mellitus (DM) type 2 is growing (1,2). Currently, some of these agents have been approved in combination with insulin. The potential for combined use with insulin has garnered increasing attention due to reduce side effects associated with insulin therapy and improve glycemic control. Some investigators reported that GLP-1 analogue combined with insulin reduces HbA1c and weight with low risk of hypoglycemia and high treatment satisfaction (3). However, their duration of treatment was short time with less than a mean of 3.0 years and the alterations of chronic diabetic complications by combination with incretin-based and insulin therapies are not known.

We evaluated the long effects of adding incretin-based therapy (DPP-4 inhibitors or GLP-1 analogues) to insulin therapy on glycated hemoglobin (HbA1c) as glycemic control, body mass index (BMI), blood pressure (BP), insulin dosage, frequency of hypoglycemia, and chronic diabetic complications for 5 years-treatments.

DETAILED DESCRIPTION:
Patients were treated with diet, exercise, and/or oral conventional pharmacotherapy combined with insulin. Oral conventional pharmacotherapy consisted of α-glycosidase inhibitors (α-GI), sulfonylurea (SU), biguanide (BG), thiazolidinedione (TZD), or combinations of these agents. Insulin therapy consisted of subcutaneous injections of long-acting insulin analogues prior to sleep and bolus subcutaneous injections of rapid-acting insulin analogues in multiple daily injections, or subcutaneous injections of mixed insulin analogues twice a day. In spite of the treatments, when the physician in charge judged that their values of HbA1c were inappropriate, the physician added the pharmacotherapy combined the insulin to incretin-based therapy. 2.3.2. For ethical reasons, patients were treated with various anti-hypertensive, anti-diabetic, anti-dyslipidemia and/or anti-hypercoagulation agents during the course of the study by the patients' own doctors as a part of continuing standard medical care. As to the drugs that have been used for the treatment of other disorders and its complication since the time before the study, the content should not be changed during the study in principle unless the complication is cured. If any new complication occurs during the study period, an appropriate treatment is given by the judgment of investigator.

ELIGIBILITY:
Inclusion Criteria:

After a detailed baseline examination, 500 Japanese subjects with type 2 diabetes were followed up for all-cause mortality and morbidity. All participants visited our clinic regularly. All patients were fully informed about the purposes and procedures for the study and provided oral consent at enrolment.

Exclusion Criteria:

Patients participating in other clinical study. Other than the above, patients judged inappropriate as the subjects of this study by the investigator.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Death | Duration varied between individual patients and was as the period of time after treatment with incretin-based therapy combined with insulin.
  The cause of death was determined by attending doctor or was assessed by interviewing the family.

SECONDARY OUTCOMES:
HbA1c | Average time requires 5 years
  Duration varied between individual patients and was as the period of time until after treatment with incretin-based therapy combined with insulin.
BMI | Average time requires 5 years
  BMI was calculated from body weight and height for at baseline and every 3 to 6 months throughout the study.
Blood pressure | Average time requires 5 years
  Participants were examined using the same methods reported previously (4). Briefly, BP was measured in the clinic and at home on waking in the morning at trough by the same methods included device, device validation, observer, number of measurements, conditions, posture and cuffs described previously (4). Namely, clinic BP (CBP) was measured once in each clinic visit. Home BP (HBP) was measured every day in the morning within 10 minutes after awakening in the sitting position.
Insulin dose | Average time requires 5 years
  Patients were treated with insulin analogues using MDI, or twice-daily injections. The dose was estimated by medical records.
Hypoglycemia | Average time requires 5 yearsinsulin.
  Patients were treated with insulin analogues using MDI, or twice-daily injections. The dose was estimated by medical records.
Hypoglycemia | Average time requires 5 years
  Hypoglycemia and the number of time per day were assessed by medical examination owing to interview.
Microvascular complications including renal anemia | Average time requires 5 years
  They were assessment by the method mentioned above. As renal anemia, serum hemoglobin (Hb) was measured by cyanmet-hemoglobin method using commercial reagent.
Macrovasular complications | Average time requires 5 years
  They were confirmed by medical history, including contents of treatment. New or worsened (recurrent) events were defined based on clinical manifestations and treatment throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital
Locations (1):
- Nagaoka Red Cross Hospital, Nagaoka, Niigata, Japan

REFERENCES:
- [Result] 1. Rizos EC, Ntzani EE, Papanas N, Tsimihodimos V, Mitrogianni Z, Maltezos E, Elisaf MS. Combination therapies of DPP4 Inhibitors and GLP1 analogues with insulin in type 2 diabetic patients: A systematic review. Curr Vasc Pharmacol. 2012 Jun 22. [Epub ahead of print] 2. Jendle J, Martin SA, Milicevic Z. Insulin and GLP-1 analog combinations in type 2 diabetes mellitus: a critical review. Expert Opin Investig Drugs. 2012 Jul 16. [Epub ahead of print] 3. Lind M, Jendle J, Torffvit O, Lager I. Glucagon-like peptide 1 (GLP-1) analogue combined with insulin reduces HbA1c and weight with low risk of hypoglycemia and high treatment satisfaction. Prim Care Diabetes. 2012; 6: 41-46. 4. Kamoi K, Miyakoshi M, Soda S, Kaneko S, Nakagawa O. Usefulness of home blood pressure measurement in the morning in type 2 diabetic patients. Diabetes Care 2002; 25: 2218-2223.